CLINICAL TRIAL: NCT07082855
Title: A Multicenter, Double-Blind, Randomized Controlled Clinical Study of Minocycline for the Treatment of Retinitis Pigmentosa
Brief Title: A Multicenter, Randomized, Double-Blind, Controlled Clinical Study of Minocycline for the Treatment of Retinitis Pigmentosa
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Liang Dan, Zhongshan Ophthalmic Center, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRP
Record Dates: First submitted 2025-07-15; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Retinitis Pigmentosa; Inherited Retinal Dystrophy; Retina Disorder
Keywords: Retinitis Pigmentosa; Minocycline; ERG; Inherited Retinal Dystrophy
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Diseases; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Minocycline 100mg (Experimental): Capsules Minocycline 100mg po once in the morning and placebo 100mg po once in the evening for 12 months
  Interventions: Drug: Minocycline 100mg
- Minocycline 200mg (Experimental): Capsules Minocycline 100mg po twice a day for 12 months
  Interventions: Drug: Minocycline 200mg
- Placebo (Placebo Comparator): Capsules placebo 100mg po twice a day for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline 100mg — Capsules Minocycline 100mg po per day and placebo 100mg po per day for 12 months
  Other Names: MRP intervention 1
  Arms: Minocycline 100mg
Drug: Minocycline 200mg — Capsules Minocycline 100mg po twice a day for 12 months
  Other Names: MRP intervention 2
  Arms: Minocycline 200mg
Drug: Placebo — Capsules placebo 100mg po twice a day for 12 months
  Other Names: MRP control
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized controlled clinical trial to get high - level evidence on minocycline's efficacy and safety（100mg/d, 200mg/d) for Retinitis pigmentosa and to find the optimal treatment dose.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a major blinding eye disease, with a global prevalence of 1/9000-1/850. It's estimated that over 1.5 million Chinese people may have RP. Its typical clinical features are night blindness and progressive tunnel vision. In the disease's end stage, total loss of peripheral and central vision may occur, accounting for about 20% of all blinding causes. The main characteristic of RP is the progressive apoptosis of retinal photoreceptor cells, which leads to gradually worsening night blindness, concentric visual field constriction, and decreased visual acuity, among other visual function impairments.

The core of RP treatment is to slow down the progression of visual impairment and delay disease advancement. However, currently there are no effective clinical methods or recommended medications to control or slow RP's progression. In recent years, advanced therapies like gene therapy and stem cell treatments have been tried for RP but are still far from clinical application due to technical challenges. So, there's an urgent need for more accessible, widely applicable, and economical treatments.

RP has a complex and poorly understood etiology. Microglia, key resident macrophages in the central nervous system, when activated, can promote neurodegenerative diseases like RP. Suppressing this activation may slow disease progression. Minocycline, a tetracycline antibiotic with anti-inflammatory and immunomodulatory effects, can cross the blood - brain barrier and protect neurons by inhibiting microglial activation. It's been studied for treating neurodegenerative diseases such as Alzheimer's and Huntington's disease. A randomized controlled trial published in The New England Journal of Medicine in 2017 found that 6 months of 200mg daily minocycline for clinically isolated syndrome patients reduced their conversion rate to multiple sclerosis, showing minocycline's potential in neurodegenerative disease treatment. Safety studies indicate no antibiotic resistance after 36 months of 200mg daily minocycline used in geographic atrophy in age-related macular degeneration.

Our team completed a pilot study on minocycline for RP. The results showed that 12 months of 100mg daily minocycline improved RP patients' visual function with good tolerability.

Based on this, we plan a multicenter, randomized, double-blind, controlled clinical trial to get high - level evidence on minocycline's efficacy and safety for RP.

ELIGIBILITY:
Inclusion Criteria:

* Age should be between 18 and 60 years old.
* Clinically diagnosed with retinitis pigmentosa, characterized by reduced electroretinogram (ERG) responses and constricted visual fields.
* In at least one eye, the amplitude of the 30Hz flicker ERG under photopic conditions should not be lower than 0 microvolts.
* The best-corrected visual acuity (BCVA, ETDRS) in both eyes should not be lower than 0.

Exclusion Criteria:

* Allergic to tetracycline antibiotics.
* Pregnant or breastfeeding.
* Syndromic retinitis pigmentosa.
* Currently taking tetracycline antibiotics or any medications that may have adverse interactions with minocycline.
* Currently participating in or having participated in another investigational study within the past 6 months.
* Presence of other ocular diseases, including glaucoma, uveitis, age-related macular degeneration, diabetic retinopathy, etc.
* History of ocular surgical intervention.
* History of uncontrolled severe comorbid conditions, such as renal disease, liver disease, autoimmune disease, thyroid dysfunction, psychiatric disorders, or idiopathic intracranial hypertension.
* Inability of the participant to comply with the study-required procedures, such as epilepsy, inability to fixate, or allergy to fluorescein. Inability to understand the content of the study, sign the informed consent form, or comply with the study procedures or follow-up visits.
* Inability to swallow capsules.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The change of ERG | 12 months
  The proportion of patients in the group who showed an increase in the amplitude of the light-adapted 30Hz flicker ERG response at 12 months post-treatment compared to baseline.

SECONDARY OUTCOMES:
The change of BCVA | 12 months
  The proportion of patients in this group showing an increase from baseline at month 12 of treatment.
The change of VF | 12 months
  The proportion of patients in this group showing an increase from baseline at month 12 of treatment.
The change of color vision | 12 months
  The proportion of patients in this group showing an increase from baseline at month 12 of treatment.
The change of microperimetry | 12 months
  The proportion of patients in this group showing an increase from baseline at month 12 of treatment.
The change of contrast sensitivity | 12 months
  The proportion of patients in this group showing an increase from baseline at month 12 of treatment.
The change of OCT | 12 months
  The proportion of patients in this group showing an increase from baseline at month 12 of treatment.
The change of NEI-VFQ-25 | 12 months
  The proportion of patients in this group showing an increase from baseline at month 12 of treatment.
The change of other ERG amplitude | 12 months
  The proportion of improvement in amplitude in light-adapted 3.0Hz ERG, dark-adapted 0.01Hz ERG and dark-adapted 3.0Hz ERG from baseline at month 12 of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No